CLINICAL TRIAL: NCT01192698
Title: Intravenous Interferon During the Anhepatic Phase of Liver Transplantation and Prevention of Recurrence of Hepatitis C Virus
Brief Title: Intravenous Interferon During Liver Transplant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: American College of Gastroenterology (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 04-05-09A
Record Dates: First submitted 2010-08-30; First posted 2010-09-01 (Estimated); Results first posted 2017-08-07 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2017-07

CONDITIONS: Hepatitis C; Cirrhosis
Keywords: cirrhosis; hepatitis C
MeSH Terms: conditions — Hepatitis C; Fibrosis | interventions — Interferons

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IV interferon (Experimental): IV interferon oral ribavirin
  Interventions: Drug: IV interferon
- Standard of care (No Intervention): standard of care

INTERVENTIONS:
Drug: IV interferon — IV interferon 5MU during anhepatic phase
  Arms: IV interferon

SUMMARY:
The main goal of this study is to prevent liver allograft infection with Hepatitis C virus in hepatitis C positive patients undergoing liver transplantation. The hypothesis is that patients who receive ribavirin immediately before transplant and intravenous interferon alfa 2b during the anhepatic phase(while the liver is removed)will have sustained virologic response post liver transplant.

DETAILED DESCRIPTION:
The study is evaluating intravenous interferon given during the anhepatic phase of lvier transplant. Ribavirin was given as well. Serial measurements for HCV RNA were determined 12, 24 72, 96 hrs and 4 weeks after liver transplant.

ELIGIBILITY:
Inclusion Criteria:

* liver transplant for hepatitis c

Exclusion Criteria:

* allergy to interferon

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2009-10; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark W Russo, MD, MPH, Principal Investigator — Wake Forest University Health Sciences

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- no Treatment: standard of care
Period: Overall Study
Arm/Group | IV Interferon | no Treatment
Started | 10 | 5
Completed | 10 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- IV Interferon: IV interferon oral ribavirin
  Aims The purpose of this study was to determine the safety and effect of intravenous interferon (IFN) during the anhepatic phase of LT on hepatitis C viral load. Methods Fifteen consecutive subjects undergoing liver transplant for hepatitis C cirrhosis were enrolled in the study, ten of which received study drug and five subjects served as controls. Cases received weight-based ribavirin and subcutaneous IFN at time of incision followed by intravenous IFN at the start of the anhepatic phase.
- no Treatment: standard of care for liver transplant
- Total: Total of all reporting groups
Arm/Group | IV Interferon | no Treatment | Total
Number analyzed (Participants) | 10 | 5 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 5 | 15
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 57 [49 to 64] | 55.8 [49 to 63] | 56.4 [49 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 10 | 4 | 14
Region of Enrollment [Number; unit: participants]
  United States | 10 | 5 | 15

OUTCOME MEASURES:

1. Primary Outcome: HCV RNA Result
Description: Will measure mean HCV RNA levels 4 weeks after liver transplant
Time Frame: 4 weeks after liver transplant
Measure: Mean (Standard Deviation); unit: IU/ml
Arm/Group | IV Interferon | no Treatment
Number analyzed (Participants) | 10 | 5
IU/ml | 924,082 (53,000) | 3,731,749 (64,000)

ADVERSE EVENTS:
Arm/Group | IV Interferon | no Treatment
Serious Adverse Events (participants affected / at risk) | 3/10 | 0/5
Other Adverse Events (participants affected / at risk) | 1/10 | 0/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IV Interferon (N=10) | no Treatment (N=5)
Flash pulmonary edema (Cardiac disorders) | 1 (1) | 0 (0) — Flash pulmonary edema occurred during liver transplant surgery
Acute cellular rejection (Immune system disorders) | 1 (1) | 0 (0) — Liver biopsy showed acute cellular rejection 1 week post transplant. The treating physician 's assessment is the acute rejection was most likely due to a low prograf level.
Increased leukopenia requiring administration of granulocyte colony stimulating factor (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IV Interferon (N=10) | no Treatment (N=5)
pulmonary edema (General disorders) | 1 (1) | 0 (0) — pulmonary edema

LIMITATIONS AND CAVEATS:
small sample size short duration of treatment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No